CLINICAL TRIAL: NCT07095803
Title: Ivonescimab (PD-1/VEGF Bispecific Antibody) Plus Radiofrequency Ablation for Multiple Advanced Tumors After PD-1 Therapy Failure: A Multicohort, Multicenter, Single-Arm Phase II Study
Brief Title: Ivonescimab (PD-1/VEGF Bispecific Antibody) Plus Radiofrequency Ablation for Multiple Advanced Tumors After PD-1 Therapy Failure
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sheng Zhang (Other)
Responsible Party: Sponsor-Investigator, Sheng Zhang, Prof., Fudan University
Organization: Fudan University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK112-US-02
Record Dates: First submitted 2025-07-15; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Multiple Advanced Tumors After PD-1 Therapy Failure
Keywords: Radiofrequency Ablation; Ivonescimab; Immunotherapy; Advanced Tumors
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental): Patients with advanced tumors who had been evaluated as effective on PD1 or PD1 combined with targeted therapy (CR,PR, or SD for more than 6 months on PD1 therapy) and then progressed on PD1 therapy or progressed less than 3 months after drug withdrawal;
  Interventions: Drug: Ivonescimab (20mg/kg Q3W); Procedure: radiofrequency ablation
- 2 (Experimental): Patients with advanced tumors who had been evaluated as having a response to PD1 or PD1 combined targeted therapy (CR,PR, or SD for more than 6 months on PD1 therapy) and then progressed more than 3 months after drug withdrawal.
  Interventions: Drug: Ivonescimab (20mg/kg Q3W); Procedure: radiofrequency ablation
- 3 (Experimental): Patients with advanced tumors who failed to respond to PD1 or PD1 combined with targeted therapy (the effect of PD1 therapy was PD or SD < 6 months).
  Interventions: Drug: Ivonescimab (20mg/kg Q3W); Procedure: radiofrequency ablation

INTERVENTIONS:
Drug: Ivonescimab (20mg/kg Q3W) — Patients received intravenous everciximab (20mg/kg Q3W) within 1 week before and after radiofrequency ablation.
Procedure: radiofrequency ablation — Patients received radiofrequency treatment for less than three lesions.

SUMMARY:
The goal of this clinical trial is to learn if the combination of radiofrequency ablation (RFA) and Ivonescimab (PD-1/VEGF Bispecific Antibody) works to could reverse PD-1/PD-L1 resistance in patients with advanced tumors. It will also learn about the safety of this combination. The main questions it aims to answer are:

Does the combination of RFA and Ivonescimab increase the objective response rate (ORR) of participants? What medical problems do participants have when taking the combination? Will the combination influence the progression-free survival time (PFS) and overall survival time and quality of life (QoL) of participants?

Participants will:

Patients received RGA treatment for less than three lesions. Patients were treated with Ivonescimab (20mg/kg Q3W, every 3 weeks) within 1 week before and after radiofrequency treatment until disease progression or intolerable toxicity occurred, or Ivonescimab was used for 2 years. Treatment effects will be evaluated every 9 weeks for 1 year and every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily provide written informed consent
* Age ≥18 years old
* Histologically and/or cytologically confirmed advanced tumors as assessed by imaging or ultrasound
* ECOG score: 0-2
* At least one measurable lesion (according to RECIST criteria, the major diameter of non-lymph node lesions on CT scan ≥10 mm, and the minor diameter of lymph node lesions on CT scan ≥15 mm); There are other lesions that can be treated with radiofrequency
* Blood routine: Absolute Neutrophil Count (ANC) 1.5×10^9/L, Platelet (PLT) ≥70×10^9/L, Hemoglobin (HGB) ≥80g/L
* Liver function: serum Total Bilirubin (TBIL) ≤1.5× Upper Limit of Normal Value (ULN); Alanine Aminotransferase (ALT) and Aspartate Transferase (AST) ≤3×ULN, and AST and ALT ≤5.0 ULN in patients with liver metastasis; Serum albumin ≥28 g/L
* Renal function: serum Creatinine (Cr) ≤1.5×ULN, or creatinine clearance ≥50 mL/mi (using the standard Cockcroft-Gault formula) 9. Coagulation: International Normalized Ratio (INR) ≤1.5 /PT≤1.5×ULN, aPTT≤1.5×ULN
* Estimated survival time ≥3 months
* Use of a medically approved contraceptive method is required during the study treatment period and for at least 120 days after the end of the study, and sperm donation or cryopreservation for fertilization and reproduction is not permitted during this period
* Ability to adhere to study access schedules and other protocol requirements

Exclusion Criteria:

* Subjects with any severe and/or uncontrolled illness. These include:

  1. poor blood pressure control (systolic blood pressure ≥150 MMHG or diastolic blood pressure ≥100 MMHG); Poorly controlled diabetes (fasting blood glucose [FBG] > 10mmol/L);
  2. with ≥ grade 2 myocardial ischemia or myocardial infarction, arrhythmia (QTc≥470ms), and ≥ grade 2 congestive heart failure (New York Heart Association [NYHA] classification); And 3) severe active or uncontrolled infections (≥CTCAE grade 2 infection) requiring systemic antibacterial, antifungal, or antiviral therapy, including pulmonary tuberculosis infection.

  4) patients with a history of active tuberculosis; 5) If it is not controlled, ascites, pericardial effusion and pleural effusion still need repeated drainage
* Active hepatitis (transaminase did not meet the inclusion criteria, hepatitis B reference: HBV DNA≥2000 IU/ml or ≥104 copies /ml; Hepatitis C reference: HCV RNA≥2000 IU/ml or ≥104 copies /ml; After nucleotide antiviral therapy, those below the above criteria can be enrolled). Chronic hepatitis B virus carriers with HBV DNA < 104 IU/ml could only be enrolled if they received antiviral therapy at the same time during the trial
* A history of immunodeficiency, including HIV infection or other acquired or congenital immunodeficiency diseases
* Active autoimmune disease requiring systemic treatment within 2 years before the initiation of treatment, or autoimmune disease with potential recurrence or planned treatment as judged by the investigator; Exceptions include skin diseases that do not require systemic treatment (e.g., vitiligo, alopecia, psoriasis, or eczema); Hypothyroidism due to autoimmune thyroiditis requires only stable doses of hormone replacement therapy. Well-controlled type I diabetes; Subjects who have had complete remission of childhood asthma without any intervention in adulthood; The investigator judged that the disease would not recur in the absence of an external trigger
* Received non-specific immunomodulatory therapy (such as interleukin, interferon, thymosin, etc., excluding IL-11 for thrombocytopenia) within 2 weeks before the first dose
* Subjects required systemic treatment with corticosteroids (>10mg prednisone equivalent per day) or other immunosuppressive drugs within 14 days prior to study initiation. Subjects allowed topical, ocular, intra-articular, intranasal, and inhaled corticosteroids. Physiological alternative doses of systemic corticosteroids are allowed. Allowing short-term use of corticosteroids for prevention (e.g., contrast allergy) or treatment of non-autoimmune conditions (e.g., delayed hypersensitivity from contact allergens)
* Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation
* Known presence, leptomeningeal metastasis, spinal cord metastasis or compression
* History of abdominal fistula or gastrointestinal perforation related to anti-VEGF therapy; Esophagogastric varices, severe ulcers, unhealed wounds, gastrointestinal perforation, abdominal fistula, gastrointestinal obstruction, intra-abdominal abscess, acute gastrointestinal bleeding, extensive bowel resection (partial colectomy or extensive small bowel resection with chronic diarrhea), Crohn's disease, ulcerative colitis, or long-term chronic diarrhea within 6 months before the first administration of the drug
* Unhealed or poorly healed wounds or active ulcers
* Failure to resolve toxicity from previous antineoplastic therapy, defined as failure to return to NCI CTCAE version 5.0 grade 0 or 1
* Patients who underwent major surgical treatment, open biopsy, or significant traumatic injury within 28 days before the start of study treatment; Or have a wound or fracture that has not healed for a long time
* Severe hypersensitivity reaction after using monoclonal antibody; Those who were known to be allergic to the active ingredients or excipients of the study
* Are participating or have participated in other clinical investigators within 4 weeks before study initiation
* Have received a live vaccine within 30 days before the first dose, or plan to receive a live vaccine during the study
* Patients with a history of severe allergy
* At risk of bleeding, or coagulopathy, or receiving thrombolytic therapy
* Persons with a history of psychotropic drug abuse and inability to quit or mental disorders
* Subjects who, in the investigator's judgment, had a concomitant medical condition that seriously jeopardized the safety of the subjects or interfered with the completion of the study, or who were deemed to be ineligible for enrollment for any other reason. A clear history of a previous neurological and mental disorder, such as dementia, epilepsy, or seizure prone
* The presence of concomitant diseases (such as severe diabetes mellitus, thyroid disease, and psychosis), or serious and/or unstable medical, psychiatric, or other conditions (including laboratory abnormalities) that, in the judgment of the investigators, seriously compromise the safety of the subjects or prevent the subjects from completing the study, or the presence of serious and/or unstable medical, psychiatric, or other conditions (including laboratory abnormalities) that affect the safety of the patients or affect the informed consent of the patients; Or the presence of any psychological, family, sociological or geographical factors that affect the study protocol and follow-up plan
* The investigator decided that he was not suitable to participate in the trial for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who achieved CR or PR according to RECIST V.1.1 criteria. | Efficacy was assessed every 9 weeks for 1 year and every 12 weeks thereafter (assessed up to 3 years).
  Objective Response Rate (ORR)

SECONDARY OUTCOMES:
Time from treatment start to progression by RECIST V.1.1. | From date of treatment until the date of first documented progression, assessed up to 100 months.
  Progression-free survival(PFS)
Time from treatment start to death of participants. | From date of treatment until the date of death from any cause, whichever came first, assessed up to 100 months.
  Overall Survival(OS)
Type, incidence, severity, onset and end time of adverse events (AE) evaluated according by the version 5.0 of NCI-CTCAE. | Began at 30 days (±7 days) after the last study treatment to 1 year.
  Evaluation of safety
Scores based on the assessment of FACT-P, version 4. | Assessments were performed every 6 weeks during the screening period and during treatment (assessed up to 1 year).
  Quality of Life (QoL) among participants. Scores based on the assessment of FACT-P, version 4, range from 0-156 points. Higher scores mean a better outcome.

IPD SHARING:
Plan to Share IPD: No